CLINICAL TRIAL: NCT05350501
Title: A Phase 2 Trial of EO2040, a miCrobiaL-derived Peptide therApeUtic Vaccine, in Combination With Nivolumab, for Treatment of Patients With ctDNA-dEfined Minimal Residual Disease of CRC Stage II, III, or IV After Curative Therapy
Brief Title: EO2040 in Combination With Nivolumab, for Treatment of Patients With Minimal Residual Disease of Colorectal Cancer
Acronym: CLAUDE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: the study recruitment is significantly behind expectations as only one single patient has started treatment
Sponsor: Enterome (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EOCRC1-22
Record Dates: First submitted 2022-04-06; First posted 2022-04-28 (Actual); Results first posted 2024-12-19 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patients With Minimal Residual Disease of Colorectal Cancer (Experimental): Patients With Circulating Tumor DNA-defined Minimal Residual Disease of Colorectal Cancer Stage II, III, or IV After Completion of Curative Therapy
  Interventions: Drug: EO2040

INTERVENTIONS:
Drug: EO2040 — EO2040, is a therapeutic peptide vaccine composed of two microbial-derived peptides mimicking cytotoxic T cell (CD8+ T cell) epitopes from the Tumor Associated Antigens (TAAs) combined with the helper peptide (CD4+ T cell epitope) Universal Cancer Peptide 2 (UCP2).
  The peptide mix EO2040, i.e. drug product (DP), will be emulsified with the adjuvant Montanide.
  EO2040 will be given in combination with nivolumab, which is an anti-PD1. Nivolumab is approved for use for the treatment of multiple cancer types, including subtypes of CRC (mismatch repair deficient or microsatellite instability-high metastatic disease after prior treatment). However, it is not currently approved for ctDNA defined MRD of CRC.
  Other Names: Nivolumab

SUMMARY:
The current study will evaluate the microbiome-derived therapeutic vaccine EO2040 in combination with nivolumab in patients with circulating tumor DNA-defined Minimal Residual Disease (MRD) of colorectal cancer stage II, III, or IV after completion of standard curative therapy.

DETAILED DESCRIPTION:
The microbiome-derived therapeutic vaccine concept utilized in conjunction with anti-Programmed cell Death protein 1 (PD1) blockade is an innovative option for testing of a rational immunotherapy in colorectal cancer. The concept as such, including the combination with nivolumab, has already been tested in the clinical setting (i.e. in recurrent glioblastoma and adrenal tumors) and shown to be well tolerated.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to receive study treatment, a patient must meet all the criteria below:

1. Provided written informed consent prior to any study-related procedures .
2. Histological confirmation of colorectal cancer.
3. Post R0-resection of stages II, III, or IV CRC and completion of all planned standard of care adjuvant therapies.
4. Presence of minimal residual disease as defined by a positive ctDNA assay after completion of all planned standard of care therapies.
5. Age ≥ 18 years old.
6. Human leukocyte antigen (HLA)-A2 positive.
7. No evidence of radiographic disease
8. Predefined performance status
9. Female patients of childbearing potential must have a negative serum pregnancy test within 72 hours prior to randomization.
10. Considering the embryofetal toxicity of the immune checkpoint inhibitor (ICI) shown in animals' models, recommendations for contraception must be followed.
11. Patients willing and able to comply with the scheduled visits, treatment plan, laboratory tests, and other study procedures indicated in the protocol.

Exclusion Criteria:

Patients who meet any of the following criteria will not be eligible to participate in the study:

1. Patients treated with dexamethasone > 2 mg/day or equivalent .
2. Patients treated with radiotherapy within 12 weeks, and cytotoxic chemotherapy therapy within 28 days (or 5 half lives of the compound(s) administered if longer) before study treatment start.
3. Patients with persistent Grade ≥ 2 toxicities (according to NCI-CTCAE v5.0). Toxicities must be resolved for at least 2 weeks to Grade 1 or less. However, alopecia, neuropathy, and other persisting toxicities not constituting a safety risk based on Investigator's judgment are acceptable.
4. Patients who have received any prior treatment with compounds targeting PD1, PD-L1, Cytotoxic T-lymphocyte-associated Antigen 4 (CTLA-4), or similar compounds where general resistance against therapeutic vaccination approaches might have developed.
5. Patients with defined abnormal laboratory values:
6. Patients with presence of other concomitant active, invasive malignancies .
7. Patients with clinically significant active infection, cardiac disease, significant medical or psychiatric disease/condition that, in the opinion of the Investigator, would interfere with the interpretation of patient safety or study results or that would prohibit the understanding or rendering of informed consent
8. Patients with suspected autoimmune or active autoimmune disorder or known history of an autoimmune neurologic condition (e.g., Guillain-Barré syndrome)..
9. Patients with a history of solid organ transplantation or allogeneic hematopoietic stem cell transplantation.
10. Patients with a history or known presence of tuberculosis.
11. Pregnant and breastfeeding patients.
12. Patients with a history or presence of human immunodeficiency virus (HIV) and/or active hepatitis B virus (HBV)/hepatitis C virus (HCV).
13. Patients who have received live or attenuated vaccine therapy used for prevention of infectious diseases including seasonal (influenza) vaccinations within 4 weeks of the first dose of study drug.
14. Patients with a history of hypersensitivity to any excipient, or active substance, present in the pharmaceutical forms of applicable study treatments.
15. Patients under treatment with immunostimulatory or immunosuppressive medications, including herbal remedies, or herbal remedies known to potentially interfere with major organ function.
16. Patients who have received treatment with any other investigational agent, or participation in another clinical trial

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2024-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Fagerberg, MD, Study Director — Enterome
Locations (1):
- MD Anderson, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Minimal Residual Disease of Colorectal Cancer: Patients With Circulating Tumor DNA-defined Minimal Residual Disease of Colorectal Cancer Stage II, III, or IV After Completion of Curative Therapy
  EO2040: EO2040, is a therapeutic peptide vaccine composed of two microbial-derived peptides mimicking cytotoxic T cell (CD8+ T cell) epitopes from the Tumor Associated Antigens (TAAs) combined with the helper peptide (CD4+ T cell epitope) Universal Cancer Peptide 2 (UCP2).
  The peptide mix EO2040, i.e. drug product (DP), will be emulsified with the adjuvant Montanide.
  EO2040 will be given in combination with nivolumab, which is an anti-PD1. Nivolumab is approved for use for the treatment of multiple cancer types, including subtypes of CRC (mismatch repair deficient or microsatellite instability-high metastatic disease after prior treatment). However, it is not currently approved for ctDNA defined MRD of CRC.
Period: Overall Study
Arm/Group | Patients With Minimal Residual Disease of Colorectal Cancer
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 1
Arm/Group | Patients With Minimal Residual Disease of Colorectal Cancer
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Median (Standard Deviation); unit: years] | 42 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1
BMI [Number; unit: kg/m2] | 39

OUTCOME MEASURES:

1. Primary Outcome: Response to Treatment at 6 Months
Description: Percentage of patients with ctDNA clearance and no radiographic evidence of recurrence
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Minimal Residual Disease of Colorectal Cancer
Number analyzed (Participants) | 1
Participants | 0

2. Secondary Outcome: Treatment-Emergent Adverse Events
Description: Number and percentage of patients with Treatment-Emergent Adverse Events (TEAEs)
Time Frame: 7 months
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Minimal Residual Disease of Colorectal Cancer
Number analyzed (Participants) | 1
Participants | 1

3. Secondary Outcome: Serious Adverse Events
Description: Number and percentage of patients with Serious Adverse Events (SAEs )
Time Frame: 7 months
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Minimal Residual Disease of Colorectal Cancer
Number analyzed (Participants) | 1
Participants | 1

4. Secondary Outcome: NCI-CTCAE Grading
Description: Number and percentage of patients with at least one NCI-CTCAE v5.0 grade increase or decrease
Time Frame: 7 months
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Minimal Residual Disease of Colorectal Cancer
Number analyzed (Participants) | 1
Participants | 1

5. Secondary Outcome: Response to Therapy at 3 Months
Description: Percentage of patients with ctDNA clearance and no radiographic evidence of recurrence
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Minimal Residual Disease of Colorectal Cancer
Number analyzed (Participants) | 1
Participants | 0

6. Secondary Outcome: DIsease-free Survival
Description: Disease-free survival (DFS) defined as the time from start of study treatment to the date of first documented colorectal cancer (CRC) recurrence or death due to any cause,
Time Frame: 7 months
Measure: Number; unit: weeks
Arm/Group | Patients With Minimal Residual Disease of Colorectal Cancer
Number analyzed (Participants) | 1
weeks | 14

7. Secondary Outcome: Overall Survival
Description: Overall survival (OS), measured as the time from start of study treatment until death from any cause.
Time Frame: 7 months
Measure: Number; unit: months
Arm/Group | Patients With Minimal Residual Disease of Colorectal Cancer
Number analyzed (Participants) | 1
months | 7

8. Secondary Outcome: Immunogenicity and Cross-reactivity
Description: Percentage of patients with a positive tetramer staining in peripheral blood mononuclear cells for the two microbial-derived peptides which are part of the therapeutic vaccine EO2040.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Minimal Residual Disease of Colorectal Cancer
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Time Frame: 7 months
Description: 1
Arm/Group | Patients With Minimal Residual Disease of Colorectal Cancer
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Minimal Residual Disease of Colorectal Cancer (N=1)
Injection site reaction (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Minimal Residual Disease of Colorectal Cancer (N=1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Rash pustular (Infections and infestations) | 1 (1)
Blood thyroid stimulating hormone decreased (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-07-04): https://cdn.clinicaltrials.gov/large-docs/01/NCT05350501/Prot_003.pdf
  • Statistical Analysis Plan (2024-03-06): https://cdn.clinicaltrials.gov/large-docs/01/NCT05350501/SAP_004.pdf